CLINICAL TRIAL: NCT04989023
Title: Clinical Applications of Blood Flow Restriction and Rehabilitation Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aspetar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: F202007001
Record Dates: First submitted 2021-07-03; First posted 2021-08-04 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Knee Pain Chronic; Anterior Knee Pain Syndrome; Patellofemoral Pain Syndrome; Rotator Cuff Impingement Syndrome; Rotator Cuff Tendinosis
Keywords: Blood flow restriction training; Rotator cuff related shoulder pain; Low load resistance training
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Shoulder Impingement Syndrome; Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessment at baseline and at all follow-up sequence will be conducted by physiotherapists blinded to the group allocation and previous evaluation data of the patient. Participants will blinded to the sham-blood flow restriction application. They will informed that two different percentages of complete occlusion will be evaluated in terms of their effect in pain following low load exercise loading with blood flow restriction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blood flow restriction (BFR) with low load resistance training (knee) (Experimental): Patients will perform slow open kinetic chain (OKC) knee extension (90°-0°) (2s con, 2s ecc, metronome). A modified pain monitoring will dictate the loading to ≤5 kg with maximum of 4/10 pain. Patients will complete 4 sets (1x30, 3x15 reps) with 30 s rest in between. If the patient fails to shadow the pace of the metronome or to fully extend the knee, the load will be reduced by 0.5Kg. The patients will exercise in sitting with an inflatable cuff of 10cm width and 75cm length will be attached to the most proximal part of the lower extremity. The cuff will remain inflated (80% limb occlusion pressure) throughout the loading session. All participants will undergo a 45-min physiotherapy session, consisting of resistance training (3-4 sets, last set to volitional fatigue), core, and balance exercise. A modified pain monitoring approach will dictate the selection of exercises and the training load (maximum of 4/10 pain).
  Interventions: Other: Blood flow restriction (BFR) with low load resistance training
- Sham-Blood flow restriction (sham-BFR) with low load resistance training (knee) (Sham Comparator): Patients will perform slow open kinetic chain (OKC) knee extension (90°-0°) (2s con, 2s ecc, metronome). A modified pain monitoring will dictate the loading to ≤5 kg with maximum of 4/10 pain. Patients will complete 4 sets (1x30, 3x15 reps) with 30 s rest in between. If the patient fails to shadow the pace of the metronome or to fully extend the knee, the load will be reduced by 0.5Kg. The patients will exercise in sitting with an inflatable cuff of 10cm width and 75cm length will be attached to the most proximal part of the lower extremity. The cuff will remain inflated (enough room for two fingers between the skin and the cuff) throughout the loading session. All participants will undergo a 45-min physiotherapy session, consisting of resistance training (3-4 sets, last set to volitional fatigue), core, and balance exercise. A modified pain monitoring approach will dictate the selection of exercises and the training load (maximum of 4/10 pain).
  Interventions: Other: Blood flow restriction (BFR) with low load resistance training
- Blood flow restriction (BFR) with low load resistance training (shoulder) (Experimental): Patients will perform slow full range dumbbell biceps curls (2s con, 2s ecc, metronome).Initial load approximately set to 5% of the participants body weight. Patients will complete 4 sets of biceps curls (1x30, 3x15 reps) with 30 s rest between sets.If the patient fails to shadow the pace of the metronome or to fully flex the shoulder, the load will be reduced by 0.5Kg. The patients will exercise in standing with an inflatable cuff of 6cm width and 60cm length will be attached to the most proximal part of the limb. The cuff will remain inflated (60% of the limb complete occlusion pressure) throughout the loading session. All participants will undergo a 45-min physiotherapy session, exercises of the scapula stabilizers, resistance exercises of the rotator cuff muscles (3-4 sets, last set to volitional fatigue), and functional and shoulder proprioception. A modified pain monitoring approach will dictate the selection of exercises and the training load (maximum of 4/10 pain).
  Interventions: Other: Blood flow restriction (BFR) with low load resistance training
- Sham-Blood flow restriction (sham-BFR) with low load resistance training (shoulder) (Sham Comparator): Patients will perform slow full range dumbbell biceps curls (2s con, 2s ecc, metronome).Initial load approximately set to 5% of the participants body weight. Patients will complete 4 sets of biceps curls (1x30, 3x15 reps) with 30 s rest between sets.If the patient fails to shadow the pace of the metronome or to fully flex the shoulder, the load will be reduced by 0.5Kg. The patients will exercise in standing with an inflatable cuff of 6cm width and 60cm length will be attached to the most proximal part of the limb. The cuff will remain inflated (enough room for two fingers between the skin and the cuff) throughout the loading session. All participants will undergo a 45-min physiotherapy session, exercises of the scapula stabilizers, resistance exercises of the rotator cuff muscles (3-4 sets, last set to volitional fatigue), and functional and shoulder proprioception. A modified pain monitoring approach will dictate the selection of exercises and the training load (max of 4/10 pain).
  Interventions: Other: Blood flow restriction (BFR) with low load resistance training

INTERVENTIONS:
Other: Blood flow restriction (BFR) with low load resistance training — Combination of low load resistance exercise in the upper or lower limb with the addition of blood flow restriction or sham-blood flow restriction.
  Other Names: Sham-Blood flow restriction (sham-BFR) with low load resistance training

SUMMARY:
The study aims to evaluate the effect of low load resistance training combined with blood flow restriction or sham blood flow restriction in patients with anterior knee pain and rotator cuff related shoulder pain in a cross-over two-arm randomized, participant and assessor blinded design. More specifically, we aim to investigate the acute and short-term hypoalgesic response (by evaluating pressure pain detection thresholds) of low load exercise with blood flow restriction or sham blood flow restriction, the effect of these interventions in pain during clinical testing, and the possibility of a placebo effect.

DETAILED DESCRIPTION:
Exercise-induced hypoalgesia describes an acute reduction in pain sensitivity following exercise.The hypoalgesic response following different types of exercise (aerobic, resistance) has been widely investigated. Preliminary evidence suggests that blood flow restriction training may decrease pain in patients with musculoskeletal conditions. This effect may result from exercise alone, or from blood flow restriction and exercise in combination. However, the possibility that the effects seen are the result of the placebo effect cannot be discounted. The evidence for the hypoalgesic response (improvement in pain perception) following training with blood flow restriction in anterior knee pain, shoulder pain, and general musculoskeletal conditions, as well as the mechanism of blood flow restriction training inducing acute pain reduction, is sparse.Hence, this study aims to evaluate the effect of low load resistance training combined with blood flow restriction or sham blood flow restriction in patients with anterior knee pain and rotator cuff related shoulder pain in a cross-over two-arm randomized, participant and assessor blinded design. More specifically, we aim to investigate the acute and short-term hypoalgesic response (by evaluating pressure pain detection thresholds) of low load exercise with blood flow restriction or sham blood flow restriction, the effect of these interventions in pain during clinical testing, and the possibility of a placebo effect.

ELIGIBILITY:
Anterior Knee Pain patients We will recruit 40 male adult participants who had consulted a sports medicine physician in a primary care setting for anterior knee pain complaints. A standardized history and physical examination will be conducted by the physiotherapists of the rehabilitation department for inclusion in the study.

Inclusion criteria:

* age over 18 years,
* diagnosis of AKP confirmed by history and physical examination (with or without imaging) for more than six weeks
* non-traumatic history of pain onset
* pain at least during one of the three functional tests used as outcome measure (single-leg shallow leg squat, single-leg deep knee squat, step down)
* pain equal or greater than 3/10 on a numeric pain rating scale (at least in 2/3 functional tests)
* unobstructed knee range of motion and no pain in passive end-range knee extension

Exclusion criteria:

* BMI greater than 28
* systemic pathology including inflammatory joint disease or neoplastic disorders
* history of deep venous thrombosis
* hypertension (systolic pressure >140mmHg)
* history of endothelial dysfunction
* peripheral vascular disease
* diabetes
* knee pain referred from the spine
* history of previous neurological conditions
* any previous medical treatment including injections (past 3 months) or drug therapy (i.e., anti-inflammatory drugs the last 2 weeks)
* infection
* previous blood flow restriction training
* inability to understand written and spoken English or Arabic.

Rotator cuff related shoulder pain patients We will recruit 40 male adult participants who had consulted a sports medicine physician in a primary care setting for shoulder complaints. A standardized history and physical examination were conducted by the physiotherapists of the rehabilitation department for inclusion in the study.

Inclusion criteria:

* age over 18 years
* rotator cuff related shoulder pain for more than six weeks
* pain greater than 3/10 on a numeric pain rating scale on active abduction and/or resisted external rotation at zero degrees of shoulder abduction (assessed in standing with the arm in slight abducted position)

Exclusion criteria:

* full-thickness rotator cuff tear (positive drop-arm sign and/or radiographic or ultrasonographic evidence)
* BMI greater than 28
* previous shoulder surgery or shoulder fracture
* imaging evidence of severe shoulder osteoarthritis or tendon calcification,\
* adhesive capsulitis
* systemic pathology including inflammatory joint disease or neoplastic disorders
* restriction of passive range of motion in more than two planes
* history of deep venous thrombosis
* hypertension (systolic pressure >140mmHg)
* history of endothelial dysfunction
* peripheral vascular disease
* diabetes
* shoulder pain referred from the spine
* history of previous neurological conditions
* any previous medical treatment including injections (past 3 months) or drug therapy (i.e., anti-inflammatory drugs the last 2 weeks)
* infection
* previous BFR training
* inability to understand written and spoken English or Arabic

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pressure pain detection thresholds - PPDTs (knee) | Baseline
  Assessed using a hand-held mechanical pressure algometer (Wagner Instruments) with a 1cm2 rubber disk attached to the pressure gauge by applying the probe perpendicularly to the skin at a pressure rate increase of approximately 1kgf/sec. One assessor blinded to group allocation will obtain measurements with the patient in long sitting with both arms resting on the plinth. PPDTs assessment sites will be marked and evaluated over the most painful location on the knee (when this will be behind the patella the algometer will be placed on the center of patella), the tibialis anterior (halfway between the most superior attachment to the tibia and its tendon in the upper one third of the muscle belly, and the extensor carpi radialis (5cm distal to the lateral epicondyle). The average of the amount of pressure in kilograms of three trials will be used in the data analysis. The order of PPDTs assessment will be randomized among patients with 30 seconds intervals between assessments.
Pressure pain detection thresholds - PPDTs (knee) | 15 minutes
  Assessed using a hand-held mechanical pressure algometer (Wagner Instruments) with a 1cm2 rubber disk attached to the pressure gauge by applying the probe perpendicularly to the skin at a pressure rate increase of approximately 1kgf/sec. One assessor blinded to group allocation will obtain measurements with the patient in long sitting with both arms resting on the plinth. PPDTs assessment sites will be marked and evaluated over the most painful location on the knee (when this will be behind the patella the algometer will be placed on the center of patella), the tibialis anterior (halfway between the most superior attachment to the tibia and its tendon in the upper one third of the muscle belly, and the extensor carpi radialis (5cm distal to the lateral epicondyle). The average of the amount of pressure in kilograms of three trials will be used in the data analysis. The order of PPDTs assessment will be randomized among patients with 30 seconds intervals between assessments.
Pressure pain detection thresholds - PPDTs (knee) | 1 hour
  Assessed using a hand-held mechanical pressure algometer (Wagner Instruments) with a 1cm2 rubber disk attached to the pressure gauge by applying the probe perpendicularly to the skin at a pressure rate increase of approximately 1kgf/sec. One assessor blinded to group allocation will obtain measurements with the patient in long sitting with both arms resting on the plinth. PPDTs assessment sites will be marked and evaluated over the most painful location on the knee (when this will be behind the patella the algometer will be placed on the center of patella), the tibialis anterior (halfway between the most superior attachment to the tibia and its tendon in the upper one third of the muscle belly, and the extensor carpi radialis (5cm distal to the lateral epicondyle). The average of the amount of pressure in kilograms of three trials will be used in the data analysis. The order of PPDTs assessment will be randomized among patients with 30 seconds intervals between assessments.
Pain in clinical tests - Numeric Pain Rating Scale (NPRS) (knee) | Baseline
  Three standardized tests will be used in the study to assess anterior knee pain: a) Single-leg squat (shallow): the patient will be standing near a treatment bed with the height of the bed adjusted to be the mid-point of his thigh (halfway between the greater trochanter and popliteal crease), b) Single-leg squat (deep): the patient will be standing near a treatment bed and the height of the bed will be adjusted to the popliteal crease. The patient will be required to touch but not sit on the surface of the bed, and c) Step-down test: the patient will step down from a 20 cm high step using his injured limb in a slow and controlled manner, touching the ground, and returning to the starting position. Immediately after each test the patient will be asked to rate their pain on an 11-point numeric rating scale (NPRS) (0-10)
Pain in clinical tests - Numeric Pain Rating Scale (NPRS) (knee) | 15 minutes
  Three standardized tests will be used in the study to assess anterior knee pain: a) Single-leg squat (shallow): the patient will be standing near a treatment bed with the height of the bed adjusted to be the mid-point of his thigh (halfway between the greater trochanter and popliteal crease), b) Single-leg squat (deep): the patient will be standing near a treatment bed and the height of the bed will be adjusted to the popliteal crease. The patient will be required to touch but not sit on the surface of the bed, and c) Step-down test: the patient will step down from a 20 cm high step using his injured limb in a slow and controlled manner, touching the ground, and returning to the starting position. Immediately after each test the patient will be asked to rate their pain on an 11-point numeric rating scale (NPRS) (0-10)
Pain in clinical tests - Numeric Pain Rating Scale (NPRS) (knee) | 1 hour
  Three standardized tests will be used in the study to assess anterior knee pain: a) Single-leg squat (shallow): the patient will be standing near a treatment bed with the height of the bed adjusted to be the mid-point of his thigh (halfway between the greater trochanter and popliteal crease), b) Single-leg squat (deep): the patient will be standing near a treatment bed and the height of the bed will be adjusted to the popliteal crease. The patient will be required to touch but not sit on the surface of the bed, and c) Step-down test: the patient will step down from a 20 cm high step using his injured limb in a slow and controlled manner, touching the ground, and returning to the starting position. Immediately after each test the patient will be asked to rate their pain on an 11-point numeric rating scale (NPRS) (0-10)
Pressure pain detection thresholds - PPDTs (shoulder) | Baseline
  Assessed using a hand-held mechanical pressure algometer (Wagner Instruments) with a 1cm2 rubber disk attached to the pressure gauge by applying the probe perpendicularly to the skin at a pressure rate increase of approximately 1kgf/sec. One assessor blinded to group allocation will obtain measurements with the participants in long sitting with both arms resting on the plinth. PPDTs assessment sites will be marked and evaluated over the middle deltoid (muscle belly close to inferolateral insertion), the first interosseous muscle of the hand, and the tibialis anterior (halfway between the most superior attachment to the tibia and its tendon in the upper one third of the muscle belly). The average of the amount of pressure in kgs of 3 trials will be used in the data analysis. The order of PPDTs assessment will be randomized among patients with 30 secs intervals between assessments.
Pressure pain detection thresholds - PPDTs (shoulder) | 15 minutes
  Assessed using a hand-held mechanical pressure algometer (Wagner Instruments) with a 1cm2 rubber disk attached to the pressure gauge by applying the probe perpendicularly to the skin at a pressure rate increase of approximately 1kgf/sec. One assessor blinded to group allocation will obtain measurements with the participants in long sitting with both arms resting on the plinth. PPDTs assessment sites will be marked and evaluated over the middle deltoid (muscle belly close to inferolateral insertion), the first interosseous muscle of the hand, and the tibialis anterior (halfway between the most superior attachment to the tibia and its tendon in the upper one third of the muscle belly). The average of the amount of pressure in kgs of 3 trials will be used in the data analysis. The order of PPDTs assessment will be randomized among patients with 30 secs intervals between assessments.
Pressure pain detection thresholds - PPDTs (shoulder) | 1 hour
  Assessed using a hand-held mechanical pressure algometer (Wagner Instruments) with a 1cm2 rubber disk attached to the pressure gauge by applying the probe perpendicularly to the skin at a pressure rate increase of approximately 1kgf/sec. One assessor blinded to group allocation will obtain measurements with the participants in long sitting with both arms resting on the plinth. PPDTs assessment sites will be marked and evaluated over the middle deltoid (muscle belly close to inferolateral insertion), the first interosseous muscle of the hand, and the tibialis anterior (halfway between the most superior attachment to the tibia and its tendon in the upper one third of the muscle belly). The average of the amount of pressure in kgs of 3 trials will be used in the data analysis. The order of PPDTs assessment will be randomized among patients with 30 secs intervals between assessments.
Pain in isometric shoulder external rotation - Numeric Pain Rating Scale (NPRS) (shoulder) | Baseline
  The isometric test will be performed in a standardized standing position with feet shoulder width apart, hips and knees in slight flexion, elbow flexed to 90°, and wrist in neutral with the palm facing the midline. The test will be performed as a "make" test and will be repeated three times in a standardized sequence with a 10-second rest between repetitions. Participants before testing will practice two sub-maximal efforts to familiarize themselves with the task. Subsequently, they will be asked to build their force gradually to a maximum voluntary effort over a 5 second period, cued by the examiner with a monotonous voice "push…push…push…push…push…relax" to ensure consistent encouragement. The examiner will keep the dynamometer in place such that the transducer head will be aligned just proximal to the ulnar styloid process, matching the force exerted by the subject. The participants will rate their maximum pain in an 11-point numeric rating scale.
Pain in isometric shoulder external rotation - Numeric Pain Rating Scale (NPRS) (shoulder) | 15 minutes
  The isometric test will be performed in a standardized standing position with feet shoulder width apart, hips and knees in slight flexion, elbow flexed to 90°, and wrist in neutral with the palm facing the midline. The test will be performed as a "make" test and will be repeated three times in a standardized sequence with a 10-second rest between repetitions. Participants before testing will practice two sub-maximal efforts to familiarize themselves with the task. Subsequently, they will be asked to build their force gradually to a maximum voluntary effort over a 5 second period, cued by the examiner with a monotonous voice "push…push…push…push…push…relax" to ensure consistent encouragement. The examiner will keep the dynamometer in place such that the transducer head will be aligned just proximal to the ulnar styloid process, matching the force exerted by the subject. The participants will rate their maximum pain in an 11-point numeric rating scale.
Pain in isometric shoulder external rotation - Numeric Pain Rating Scale (NPRS) (shoulder) | 1 hour
  The isometric test will be performed in a standardized standing position with feet shoulder width apart, hips and knees in slight flexion, elbow flexed to 90°, and wrist in neutral with the palm facing the midline. The test will be performed as a "make" test and will be repeated three times in a standardized sequence with a 10-second rest between repetitions. Participants before testing will practice two sub-maximal efforts to familiarize themselves with the task. Subsequently, they will be asked to build their force gradually to a maximum voluntary effort over a 5 second period, cued by the examiner with a monotonous voice "push…push…push…push…push…relax" to ensure consistent encouragement. The examiner will keep the dynamometer in place such that the transducer head will be aligned just proximal to the ulnar styloid process, matching the force exerted by the subject. The participants will rate their maximum pain in an 11-point numeric rating scale.
Strength in isometric shoulder external rotation (shoulder) | Baseline
  The isometric test will be performed in a standardized standing position with feet shoulder width apart, hips and knees in slight flexion, elbow flexed to 90°, and wrist in neutral with the palm facing the midline. The test will be performed as a "make" test and will be repeated three times in a standardized sequence with a 10-second rest between repetitions. Participants before testing will practice two sub-maximal efforts to familiarize themselves with the task. Subsequently, they will be asked to build their force gradually to a maximum voluntary effort over a 5 second period, cued by the examiner with a monotonous voice "push…push…push…push…push…relax" to ensure consistent encouragement. The examiner will keep the dynamometer in place such that the transducer head will be aligned just proximal to the ulnar styloid process, matching the force exerted by the subject. The maximum of the three trials will be used for analyses.
Strength in isometric shoulder external rotation (shoulder) | 15 minutes
  The isometric test will be performed in a standardized standing position with feet shoulder width apart, hips and knees in slight flexion, elbow flexed to 90°, and wrist in neutral with the palm facing the midline. The test will be performed as a "make" test and will be repeated three times in a standardized sequence with a 10-second rest between repetitions. Participants before testing will practice two sub-maximal efforts to familiarize themselves with the task. Subsequently, they will be asked to build their force gradually to a maximum voluntary effort over a 5 second period, cued by the examiner with a monotonous voice "push…push…push…push…push…relax" to ensure consistent encouragement. The examiner will keep the dynamometer in place such that the transducer head will be aligned just proximal to the ulnar styloid process, matching the force exerted by the subject. The maximum of the three trials will be used for analyses.
Strength in isometric shoulder external rotation (shoulder) | 1 hour
  The isometric test will be performed in a standardized standing position with feet shoulder width apart, hips and knees in slight flexion, elbow flexed to 90°, and wrist in neutral with the palm facing the midline. The test will be performed as a "make" test and will be repeated three times in a standardized sequence with a 10-second rest between repetitions. Participants before testing will practice two sub-maximal efforts to familiarize themselves with the task. Subsequently, they will be asked to build their force gradually to a maximum voluntary effort over a 5 second period, cued by the examiner with a monotonous voice "push…push…push…push…push…relax" to ensure consistent encouragement. The examiner will keep the dynamometer in place such that the transducer head will be aligned just proximal to the ulnar styloid process, matching the force exerted by the subject. The maximum of the three trials will be used for analyses.

SECONDARY OUTCOMES:
Global rating of change scale (GROC) (both knee and shoulder) | 15 minutes
  Patient-perceived pain change using a global rating of change scale (GROC) based on a 7-point Likert scale ranging from "Much better - a very important improvement" to "Much worse - an important aggravation" (not applicable at baseline)
Global rating of change scale (GROC) (both knee and shoulder) | 1 hour
  Patient-perceived pain change using a global rating of change scale (GROC) based on a 7-point Likert scale ranging from "Much better - a very important improvement" to "Much worse - an important aggravation" (not applicable at baseline)
Rating of perceived exertion (RPE) in a modified Borg's scale (Borg CR10) | 15 minutes
  Participant's rating of perceived exertion (RPE) using a modified Borg's scale (Borg CR10) immediately following the blood flow restriction or sham-blood flow restriction exercise session. The scale has been shown to be an valid alternate tool for estimating the excretion and intensity levels during resistance training. A printed version of the modified scale will be presented to the participants and will be explained that a very hard session would have a rating ≥7 out of 10 and a rating of 10 meant they were giving maximal effort and could not exert themselves any further. Accordingly, a light session may have a rating of Borg ≤2, a moderate session may have a rating of Borg >2-<5, and a hard session may have a rating of Borg ≥5-<7.
Pain during active shoulder abduction (0 to 180°) in standing in a Numeric Pain Rating Scale (NPRS) (shoulder) | Baseline
  Patients will rate their pain during active shoulder abduction (0 to 180°) in standing in a NPRS ranging from 0 to 10
Pain during active shoulder abduction (0 to 180°) in standing in a Numeric Pain Rating Scale (NPRS) (shoulder) | 15 minutes
  Patients will rate their pain during active shoulder abduction (0 to 180°) in standing in a NPRS ranging from 0 to 10
Pain during active shoulder abduction (0 to 180°) in standing in a Numeric Pain Rating Scale (NPRS) (shoulder) | 1 hour
  Patients will rate their pain during active shoulder abduction (0 to 180°) in standing in a NPRS ranging from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Korakakis, PhD, Principal Investigator — Aspetar Orthopedic and Sports Medicine Hospital
Locations (1):
- Aspetar; Qatar Orthopaedic and Sports Medicine Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided